CLINICAL TRIAL: NCT02070510
Title: An Open-label, Single Arm, Sequential, Single Centre Trial Investigating the Influence of Oral Semaglutide (NNC0113-0217) on Pharmacokinetics of Lisinopril and Warfarin in Healthy Subjects
Brief Title: A Trial Investigating the Influence of Oral Semaglutide on the Pharmacokinetics of Lisinopril and Warfarin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4065; 2013-001087-39 (EudraCT Number); U1111-1140-3741 (Other: WHO)
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide; Lisinopril; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Victim and perpetrator compounds (Experimental): Subjects receive two different victim compounds (lisinopril and warfarin) and two different perpetrator compounds (placebo semaglutide with carrier and oral semaglutide). Each dosing occasion is separated by a 7-day wash-out period.
  Interventions: Drug: semaglutide; Drug: lisinopril; Drug: warfarin; Drug: placebo

INTERVENTIONS:
Drug: semaglutide — For oral administration once daily. Doses of 5 mg and 10 mg, respectively, will be given for 7 days followed by 20 mg administered on days 43-84.
Drug: lisinopril — For oral administration. A single dose of 20 mg is administered three times either alone or conconmitantly with a perpetrator compound (days 1, 15 and 71).
Drug: warfarin — For oral administration. A single dose of 5 mg is administered three times either alone or conconmitantly with a perpetrator compound (days 8, 22 and 78).
Drug: placebo — A single dose of SNAC is administered conconmitantly with victim compounds (days 15 and 22).

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the influence of oral semaglutide (NNC0113-0217) on the pharmacokinetics of lisinopril and warfarin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-75 years (both inclusive) at time of signing informed consent
* Body mass index 20.0-29.9 kg/m^2 (both inclusive)
* A good general health based on medical history, physical examination, and results of vital signs, electrocardiogram and laboratory safety tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods. Female of child bearing potential must use effective methods of birth control for the duration of the trial and for 5 weeks following last dose. Only highly effective methods of birth control are accepted (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices)
* History of Crohn's disease, ulcerative colitis, or other inflammatory bowel disease
* Hypertension (defined as sitting systolic blood pressure above 140 mmHg and/or diastolic blood pressure above 90 mmHg). If white-coat hypertension is suspected at the screening visit, a repeated measurement is allowed
* Any blood draw in excess of 50 mL in the past month, or donation of blood or plasma in excess of 400 mL within the 3 months preceding screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-02-27 (Actual); Primary Completion 2014-08-20 (Actual); Study Completion 2014-08-20 (Actual)

PRIMARY OUTCOMES:
Area under the S-warfarin concentration-time curve | From dosing to infinity calculated from a 0-168 hours S-warfarin concentration-time-curve based on 18 sampling time points
Area under the R-warfarin concentration-time curve | From dosing to infinity calculated from a 0-168 hours S-warfarin concentration-time-curve based on 18 sampling time points
Area under the lisinopril concentration-time curve | From dosing to infinity calculated from a 0-60 hours lisinopril concentration-time-curve based on 13 sampling time points

SECONDARY OUTCOMES:
Maximum observed S-warfarin plasma concentration | 0 to 168 hours after single dose
Maximum observed R-warfarin plasma concentration | 0 to 168 hours after single dose
Maximum observed lisinopril plasma concentration | 0 to 60 hours after single dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- [Background] Baekdal TA, Borregaard J, Hansen CW, Thomsen M, Anderson TW. Effect of Oral Semaglutide on the Pharmacokinetics of Lisinopril, Warfarin, Digoxin, and Metformin in Healthy Subjects. Clin Pharmacokinet. 2019 Sep;58(9):1193-1203. doi: 10.1007/s40262-019-00756-2. PMID 30945118
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com